CLINICAL TRIAL: NCT06298292
Title: Zero Minis - Acceptability and Tolerance Market Research
Brief Title: Acceptability/Tolerance of Protein Substitutes in Tablet Form for the Dietary Management of Rare Aminoacidopathies
Acronym: ZeroMinisMR
Status: Not yet recruiting | Type: Observational
Sponsor: metaX Institut fuer Diatetik GmbH (Industry)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ZerominisCT01
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Tyrosinemia, Type I; Tyrosinemia, Type II; Tyrosinemia, Type III; Alkaptonuria; Homocystine; Metabolic Disorder; MSUD (Maple Syrup Urine Disease)
MeSH Terms: conditions — Tyrosinemias; Alkaptonuria; Metabolic Diseases; Ketosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ZeroTP minis: Intervention: Tyrosine-free and Phenylalanine-free protein substitute in tablet form. Subjects who currently take a protein substitute for the dietary management of either tyrosinaemia I, II, III or alkaptonuria will be recruited. Subjects will take the study product for 7 days. Subjects will replace some or their entire usual protein substitute with the new product. The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute.
  Interventions: Dietary Supplement: Zero minis (range of protein substitutes in tablet form)
- ZeroMet minis: Intervention: Methionine-free and Cystine-enriched protein substitute in tablet form. Subjects who currently take a protein substitute for the dietary management of homocystinuria will be recruited. Subjects will take the study product for 7 days. Subjects will replace some or their entire usual protein substitute with the new product. The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute.
  Interventions: Dietary Supplement: Zero minis (range of protein substitutes in tablet form)
- ZeroVIL minis: Intervention: Valine-, Isoleucine- and Leucine-free protein substitute in tablet form. Subjects who currently take a protein substitute for the dietary management of MSUD will be recruited. Subjects will take the study product for 7 days. Subjects will replace some or their entire usual protein substitute with the new product. The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute.
  Interventions: Dietary Supplement: Zero minis (range of protein substitutes in tablet form)

INTERVENTIONS:
Dietary Supplement: Zero minis (range of protein substitutes in tablet form) — Intervention: range of protein substitute tablets. Subjects who currently take a protein substitute for the dietary management of either tyrosinaemias or alkaptonuria, homocystinuria, or MSUD will be recruited. Subjects will take the study product for 7 days. Daily questionnaires will be completed (ease of preparation,administration; any problems or gastrointestinal effects). Subjects will replace some or their entire usual protein substitute with the new product suitable for their diagnosed rare metabolic disease. The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute. Additional questions at the beginning and end of the study will record information on organoleptic properties, presentation and packaging of the product. Routine weekly blood samples will be collected and analysed for amino acids typically for the metabolic control of the individual specified metabolic disorders as is usual clinical practice.
  Other Names: ZeroTP minis; ZeroMet minis; ZeroVIL minis

SUMMARY:
The purpose of this prospective, observational study is to evaluate the tolerability and acceptability of Zero minis, a range of protein substitute tablets for use in the dietary management of children with either TYROSINAEMIA Type I, II, III or ALKAPTONURIA, HOMOCYSTINURIA, or MAPLE SYRUP URINE DISEASE (MSUD) over the age of 7 years.

DETAILED DESCRIPTION:
The principle treatment for children with inborn amino acid disorders is a strict low protein diet. Part of this treatment requires the administration of a protein substitute in order to meet basic protein requirements for normal growth and development. Several brands of protein substitutes for inborn amino acid disorders are already available in various presentations. However, compliance with taking protein substitutes continues to be a challenge. As a low protein diet is usually recommended for life, long term compliance is always a major concern. As a result, improving the choice in terms of product type may aid compliance.

Zero minis are a range of protein substitute tablets specifically designed for use in the dietary management of rare amino acid disorders like Tyrosinaemia type I, II, III or Alkaptonuria, Homocystinuria, and MSUD in children from ≥3 years of age onwards. Zero minis are concentrated protein substitutes containing a mixture of pure amino acids (except the amino acid(s) which can´t be metabolized) enriched with vitamins, minerals and trace elements. It is anticipated that they will be a suitable alternative choice for patients with rare metabolic disorders including: tyrosinaemia type I, II, III or alkaptonuria, homocystinuria, or MSUD, broadening the variety of protein substitutes they can choose from in order to suit their lifestyle and preferences.

This is a prospective, multicentre, observational tolerance study with 15 children with rare metabolic disorders. Subjects who are currently taking a protein substitute for the dietary management of either tyrosinaemia type I, II, III or alkaptonuria, homocystinuria, or MSUD, will be recruited for a 7-day trial taking the new ready-to-use protein substitute tablets to evaluate the tolerability and acceptability of the study products. Subjects will replace some or all of their usual protein substitute with the new product suitable for their diagnosed rare metabolic disease.

During the 7-day trial subjects or caregivers will be asked to complete a daily questionnaire recording information on:

* Usage and compliance
* Ease of use and any issues with administration
* Any gastro-intestinal side-effects.

A questionnaire will also be completed at the beginning and end of the study that will consider perceptions about taste, appearance, smell, presentation and packaging of each product; ease of administration; how it is taken; and any other problems or symptoms.

The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute.

Subjects will continue to have weekly blood tests as is routine in rare metabolic disorders. The results whilst on the study product will be compared with results whilst on their usual protein substitute.

15 children out of a patient pool with tyrosinaemia type I, II, III or alkaptonuria, homocystinuria, or MSUD will be recruited. When an appropriate subject has been identified, a study information sheet will be sent to the subject or parents/caregivers. They will be invited to request further information about the study if they wish by contacting the Lead Dietitian.

Recruitment of each patient will be by written informed consent, which will be completed by the parents/primary caregivers and taken by the Lead Dietitian. Children will also complete an assent/consent form and will receive an information sheet, if considered appropriate for their level of understanding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tyrosinaemia type I, II III or Alkaptonuria requiring a tyrosine- and phenylalanine-free protein substitute.
* Diagnosis of Homocystinuria requiring a methionine-free, cystine-enriched protein substitute.
* Diagnosis of MSUD requiring a valine-, leucine- and isoleucine-free protein substitute.
* Subjects who are already taking a protein substitute for one of the specified rare metabolic disorders and are willing to try the study product for 7 days.
* Children aged 7 years and over.
* Written informed consent obtained from parental caregiver.

Exclusion Criteria:

* Presence of serious concurrent illness
* Lead Dietitian's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any children having taken antibiotics over the previous 2 weeks leading up to the study.
* Children less than 7 years of age.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 15 children out of a patient pool with proven tyrosinaemia type I, II, III or alkaptonuria, homocystinuria, or MSUD will be recruited from two specialist metabolic centres.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Daily compliance | 7 days
  Compliance, with currently prescribed protein substitute will be assessed at the beginning of the 7-days trial. Usage and compliance with the study product will subsequently assessed daily from days 1-7 using standardised questionnaires, where patients document the the amount of consumed study product vs the prescribed doses.

SECONDARY OUTCOMES:
Treatment-Emergent tolerability | 7 days
  Gastro-intestinal side effects (including diarrhoea, constipation, bloating or abdominal distension, nausea, vomiting, burping, flatulence or regurgitation and abdominal discomfort or pain) will be assessed daily via questionnaire using the scale (none today, mild, moderate or severe / really troublesome).
Patient Acceptability | 7 days
  Acceptability (ease of use and palatability) will be assessed via questionnaire daily during the study period and at the end of the study via questionnaire .
Metabolic control | 7 days
  Weekly routine blood samples will be collected and analysed for specific amino acids typically for the metabolic control of the individual specified metabolic disorders as is usual clinical practice.
Incidence of study product emergent events. | 7 days
  All adverse events will be recorded throughout the study (as and when they occur). There is no specific time frame as the frequency of adverse events can not be predicted. But as the study product is already commercially available occurence of any adverse event is unlikely.

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Professor, Principal Investigator — Birmingham Children´s Hospital

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.